CLINICAL TRIAL: NCT04686630
Title: Relationship of Selective Voluntary Motor Control Impairment and Gait Deviations in Children With Cerebral Palsy by Simple Video-Based Analysis.
Brief Title: Investigation of Relations Between Edinburgh Visual Gait Score and Selective Motor Control for Children With CP
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Cansu Sardoğan, Candidate of MSc Physiotherapist, Yeditepe University
Other Study IDs: 20173034004
Record Dates: First submitted 2020-03-17; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy, Selective Motor Control, SCALE Test, Edinburgh Gait Score
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: Only observational study
  Interventions: Other: Video based observational gait analysis and SCALE Test

INTERVENTIONS:
Other: Video based observational gait analysis and SCALE Test — Twenty-four spastic diparesis and eighteen spastic hemiparesis cases were included in the study. Data was collected from 84 lower extremities. There were 22 female and 20 male patients aged between 4-18 years. Personal and disease-related information of 42 individuals with diplegic or hemiparetic CP were recorded by using the data collection form. Information collection form; The patient's name-surname, age, gender, height, weight, history, gestational age, birth weight, SCALE Test, GMFCS, Modified Ashworth Scale (MAS), Range of Motion (ROM), EVGS, affected side and previous surgical histories were recorded and their functional levels were determined and recorded.

SUMMARY:
Children with Cerebral Palsy have generally limited selective motor control which affects their ability to complete functional tasks Selective Motor Control has been shown to correlate with specific characteristics of gait, however in video based observational gait analysis, the sub phases of the gait cycle, which are affected by selective motor control, has not been investigated in children with Cerebral Palsy. Therefore the aim of this study was determine the relationship between Edinburgh Visual Gait Score and Selective Motor Control of the Lower Extremity test in children with cerebral palsy. Forty-two cerebral palsy children with Gross Motor Function Classification System level I-II-III and between 4-18 ages were participated for the study. After the demographic characteristics and all assessments of the patients were recorded, the gait characteristics of children were assessed by video based observational gait analysis. According to Edinburgh Visual Gait Score, phases of gait were analyzed.

Keywords: Cerebral Palsy, Selective Motor Control, Gait, Edinburgh Visual Gait Score

DETAILED DESCRIPTION:
Introduction and Purpose

Cerebral palsy (CP) is a group of permanent but non-progressive neurological disorder that emerges before, during, and after the birth. That disorder causes problems in the development of movement and posture and activity limitations. Motor disorders seen in CP are frequently accompanied by sensory and perception disorders, cognitive, communication and behavioral problems. In addition, epilepsy and secondary musculoskeletal problems are also added to this issue. CP varies according to etiology, severity and location of the disorder.

It is a form of classification defined by the Surveillance of Cerebral Palsy in Europe (SCPE). This classification method according to the clinical features of children with CP; Spastic type CP, Dyskinetic type CP, Ataxic CP and Unclassified / Other ".

In spastic CP, neurological damage to the corticospinal tract (CST) results in four interconnected neuromuscular deficiencies are shortened muscle-tendon unit, muscle weakness, spasticity and impaired selective motor control (SMC). These deficits are caused by brain damage, which disconnects with descending inhibitory and excitatory signals and consecutive changes in the motor unit, muscle fiber composition and muscle growth . These causes lead to inadequate motor functions in children with CP. More involvement of sensory-motor areas may impair motor function and proprioception. As well as, these neuromuscular deficits lead to the gait disorders which have commonly seen in children with spastic CP.

Although most of the studies have focused on spasticity and muscle weakness, recent research reveals the importance of SMC. SMC is described as the ability to isolate muscle activation in a selected pattern when a voluntary movement or posture is required.SMC skills are responsible for the movement and control of joints in agile and independent manner.

The etiology of SMC loss has not been entirely understood, but it is known that voluntary movements are provided by corticospinal ways. The corticospinal pathways undertake the task of determining the direction of movement and controlling force production for movement. The corticospinal pathways are located in the periventricular white matter (PWM). PWM injury is the most common finding in magnetic resonance imaging (MRI) of children with spastic type CP .CST are located in the PWM. Therefore, especially in children with spastic type CP, SMC failure or loss is quite common.

SMC skills of the upper extremities are considered as a basic factor for the realization of many activities such as eating, participating in daily living activities, performing self-care activities and writing. In addition, SMC can be used as an important guide in clinical interventions such as botulinum toxin treatment and selective dorsal rhizotomy. For these reasons, a detailed evaluation of the SMC is of great importance. However, it is noteworthy that studies on the evaluation of SMC are insufficient. The Selective Control Assessment of the Lower Extremity (SCALE) test, as the first scale that evaluates the lower extremity in a comprehensive manner and with the high level of evidence. The SCALE test which was developed as a clinical tool for evaluating SMC in lower extremities in children with CP, stands out compared to other selective motor control tests .It has has a high level of validity and reliability. The first instrument designed specifically to evaluate SMC ability of the upper extremity is the "Selective Control of Upper Extremity Scale (SCUES). Both measuring instruments are very useful, practical and understandable.

Recent studies have been focused on the idea that SMC will guide the treatment of physiotherapy and rehabilitation. Additionally, botulinum toxin can be used as a guide in surgical procedures. Beside the influence of weakness, short muscle-tendon unit, and spasticity in gait has been studied, the impact of impaired SMC on overall gait pattern has not been investigated.

SMC problems in children with CP affects motor activities at functional level such as crawling and walking. When SMC decreases or disappears, the synergy that occurs in the lower extremity prevents the performance of gait cycle or deteriorates the quality of gait. In the literature, the effect of SMC on gait cycle investigated with 3DGA; however, impaired SMC on the sub-phases of the gait cycle was not well defined in VBOGA.

In the literature, the effects of SMC on gait were investigated by three-dimensional gait analysis (3DGA); however, 3DGA is not widely used in every clinic and requires the expensive and complicated equipment. This makes the basis for us to conduct this study.

The Edinburgh visual gait score (EVGS) was developed for gait assessment using video recordings in children with CP. Additionally, in video based observational gait analysis, the sub-phases of the gait cycle, which are affected by SMC, has not been investigated in children with CP. Therefore, the aim of this study was to determine the relationship between EVGS and selective motor control of the lower extremity in children with CP.

Material and Method This study was conducted between July 2019 and December 2019 in the Human Motion Assessment Laboratory in Istanbul to investigate the relationship between the SMC of children with CP and the Edinburgh Visual Gait Score.

The study was approved by the Medical, Surgical and Drug Research Ethics Committee of Yeditepe University Faculty of Medicine and conducted in accordance with the Declaration of Helsinki.

3.1. Participants

Prior to the study, the families and children of all children with spastic CP were informed about the purpose of the study, all the assessments to be applied during the study and the benefits of the study; families and children who volunteered to participate in the study were signed an informed consent form that they voluntarily participated in the study.

The children with CP and their families were evaluated in terms of eligibility for the study. However, children who did not meet the inclusion criteria were excluded from the study and a total of 42 children were included in the study. Both SCALE and EVGS assessment scales were applied to the 42 children included in the study. Twenty-four spastic diparesis and eighteen spastic hemiparesis cases were included in the study. Data was collected from 84 lower extremities. There were 22 female and 20 male patients aged between 4-18 years.

Criteria for inclusion in the study:

* Children with a diagnosis of diplegic or hemiparetic CP.
* Between 4-18 years old,
* GMFCS level I-II-III,
* Can understand simple verbal commands,
* The study was conducted in children of families who accepted the study.

Criteria for exclusion from the study:

* Children who do not meet the criteria for inclusion,
* Children with ataxic and dyskinetic type CP were identified.
* Children who exhibit discordant attitudes during the assessment (crying, indignation),
* Families and children who want to quit working anywhere in the study,
* Children who could not complete the assessment were identified as.

3.2. Methods This study was planned to investigate the relationship between SMC and walking of children with CP. Personal and disease-related information of 42 individuals with diplegic or hemiparetic CP were recorded by using the data collection form. Information collection form; The patient's name-surname, age, gender, height, weight, history, gestational age, birth weight, SCALE Test, GMFCS, Modified Ashworth Scale (MAS), Range of Motion (ROM), EVGS, affected side and previous surgical histories were recorded and their functional levels were determined and recorded. The evaluations used in this context are indicated below.

Assessment Methods Selective Control Assessment of the Lower Extremity (SCALE)

The SCALE test was developed by Fowler et al. (10) to evaluate SMC of the lower extremity. It is a valid and reliable assessment method that does not require any special equipment during application. Application time is approximately 10 minutes. In addition, motion of ankle joint (S1), motion of subtalar joint (S2), motion of toes joint (S3), motion of knee joint (S4) and motion of hip joint (S5) parameters of the SCALE test were evaluated separately and bilaterally five. All evaluations are performed in the sitting position except for the hip joint. When evaluating the hip joint, the participant is in the lying position with the tested hip facing up. During the evaluation, clothing that prevents the observation of the extremities of the evaluated person is more easily removed. Joints of motion can be observed and scored more easily by using a short.

The evaluation positions for each S1, S2, S3, S4 and S5 are specified separately. The patient is asked to perform the desired movement for each joint level in approximately 3 seconds and with a specific oral tempo. The degree of SMC is determined as "normal" (2 points) if the patient could move the tested joint isolated, within at least 50% of the possible range of motion and at a physiological cadence cued orally by the therapist (e.g. "flex, extend, flex"). If any deviation in performance occurred (movement performed below 50% of the range of movement, slower, with synergistic movements), selectivity was regarded as "impaired" (1 point). The score "unable" was given, if no joint movement could be made or mass-synergy-patterns occurred. The total score is obtained by adding the score obtained from the joint levels to a maximum of 10 points for each limb. Testing procedures were standardized in regards to the assessment guidelines. All tests were carried out by the same two physiotherapists, one assessing and one assisting.

SMC of each joint movement was scored on a three-point ordinal scale. SMC was scored as in addition total SCALE score (ST) was included statistical analysis.

3.2.2.5. Video Based Observational Gait Analysis Participants and their parents were informed about the evaluation and then VBOGA was performed in order to evaluate their walking with EVGS. High resolution (HD) and high frame rate (60 frames per second) Nikon Coolpix S100 camera, SanDisk 16GB memory card and tripod stand were used for recording walking trials. The camera were located at the center of a 1m x 10m walkway. Its height was adjusted considering the pelvis height of the individuals. Individuals were asked to wear comfortable clothes, e.g.; tight shorts and athletes. In case of occluded superior anterior and superior posterior spina iliac (SIAS and SIPS), shorts were adjusted so that anatomic landmarks visually observable. All trials were obtained for bare foot walking.

The camera was placed 3m away from the middle of the walkway for video recording. Subjects were asked to walk at their normal pace and looking forward. The evaluated cycles were taken approximately 3-meter part in the middle of the 10-meter walkway. where the steps where the subjects gained closest to the normal gait and gained natural walking speed, were taken into consideration while determining the steps taken into consideration. The lower extremity, which was close to the video camera, was evaluated. The proper trial was selected via checking all videos. The video files taken for subject played and investigated slow play mode and the best ones were selected for evaluation. The events were got by investigating proper time frame using frame-by-frame play property of Adobe Premiere Pro CC 2018 video editing software.

1.1. Statistical Analysis

IBM SPSS ( Statistical Package Analyze for Social Sciences ) Statistics version 25.0 software was used for statistical analysis of the findings. The suitability of the variables to normal distribution was determined by Kolmogorov-Smirnov / Shapiro-Wilk tests. The relationships between the variables were analyzed using the Spearman correlation test as they were not suitable for normal distribution. Cohen correlation classification was used to define the strength of the correlation.The twenty three participants were above the minimum sample size needed to ensure a power of 95% confidence level.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of diplegic or hemiparetic CP.
* Between 4-18 years old,
* GMFCS level I-II-III,
* Can understand simple verbal commands,

Exclusion Criteria:

* Children who do not meet the criteria for inclusion,
* Children with ataxic and dyskinetic type CP were identified.
* Children who exhibit discordant attitudes during the assessment (crying, indignation),
* Families and children who want to quit working anywhere in the study,
* Children who could not complete the assessment were identified as.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with a diagnosis of diplegic or hemiparetic CP. Between 4-18 years old, GMFCS level I-II-III, Can understand simple verbal commands,
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Impaired lower-extremity Selective Voluntary Motor Control are noticeably related with the foot and ankle movements in swing and initial stance during walking as well as the total Edinburgh Visual Gait Score and sagittal and frontal trunk movements. | about 1 year
  Edinburgh visual gait score is a tool for assessment of the gait phases. Selective Voluntary Motor Control was assessed with the SCALE Test. The SCALE Test consists of 5 items, and each item can be scored between 0 and 2 (0 = unable, 1 = impaired, 2 =normal). For each limb, high scores (maximum score of 10) indicate the best SVMC. Addition,assess of Edinburgh Visual Gait Score (EVGS) (0=normal, 1=moderate or mild pathology, 2=severe pathology). So 0 here means the best score at EVGS.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmi Muammer, Prof. Dr., Principal Investigator — Yeditepe University; Nazif Ekin Akalan, Prof. Dr., Principal Investigator — Istanbul Kültür University
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study will be published in a scientific journal.
Supporting Information: ICF

REFERENCES:
- [Derived] Sardogan C, Muammer R, Akalan NE, Sert R, Bilgili F. Determining the relationship between the impairment of selective voluntary motor control and gait deviations in children with cerebral palsy using simple video-based analyses. Gait Posture. 2021 Oct;90:295-300. doi: 10.1016/j.gaitpost.2021.08.019. Epub 2021 Aug 26. PMID 34564001